CLINICAL TRIAL: NCT02747732
Title: A Phase II Study of the Bruton's Tyrosine Kinase Inhibitor, PCI-32765 (Ibrutinib), in Combination With Bendamustine and Rituximab (BR) for Patients With Relapsed/Refractory Aggressive B Cell Lymphomas
Brief Title: Study of Ibrutinib in Combination With Bendamustine and Rituximab for Patients With Relapsed/Refractory Aggressive BCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meirav Kedmi MD (Other Government)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Meirav Kedmi MD, Dr., Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bruton's Tyrosine_Meirav Kedmi
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Diffuse Large B Cell Lymphoma; Primary Mediastinal (Thymic) Large B-cell Lymphoma; Transformed Indolent Lymphoma; Recurrent Disease; Refractory Cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Neoplasms | interventions — Bendamustine Hydrochloride; Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm (Experimental): Therapy initiation 30 days max from screening.
  Bendamustine 90 mg/m2 IV on Days 1-2, Cycles 1-6 Rituximab 375 mg/m2 IV Day 1, Cycles 1-6; a cycle is defined as 28 days Ibrutinib, 560 mg orally, once daily, continuously starting on Cycle 1, Day 1 until disease progression, toxicity or referral for allo-SCT
  Interventions: Drug: Bendamustine 90 mg/m2 IV on Days 1-2, Cycles 1-6

INTERVENTIONS:
Drug: Bendamustine 90 mg/m2 IV on Days 1-2, Cycles 1-6 — Therapy initiation 30 days max from screening.
  Bendamustine 90 mg/m2 IV on Days 1-2, Cycles 1-6 Rituximab 375 mg/m2 IV Day 1, Cycles 1-6; a cycle is defined as 28 days Ibrutinib, 560 mg orally, once daily, continuously starting on Cycle 1, Day 1 until disease progression, toxicity or referral for allo-SCT
  Other Names: Rituximab 375 mg/m2 IV Day 1, Cycles 1-6;; Ibrutinib, 560 mg orally, once daily

SUMMARY:
This is a phase 2 study of the Bruton's Tyrosine Kinase Inhibitor, PCI-32765 (ibrutinib), in combination with bendamustine and rituximab (BR) in subjects with previously treated aggressive B cell non Hodgkin lymphoma (aB-NHL) including any subtype of diffuse large B cell lymphoma (DLBCL) primary mediastinal B cell lymphoma (PMBCL), double and triple hit DLBCL, transformed indolent lymphoma, unclassifiable aggressive B cell lymphoma between DLBCL and Burkitt lymphoma. Patients with CNS involvement (primary or secondary) will be excluded. Ibrutinib (IMBRUVICA®; PCI-32765; JNJ-54179060) is a first-in-class, potent, orally-administered covalently-binding small molecule inhibitor of Bruton's tyrosine kinase currently FDA approved for the treatment of relapsed Mantle cell lymphoma (MCL), Chronic Lymphocytic Leukemia (CLL) and waldenstrom Macroglobulinemia (WM).It is under constant investigation for the treatment of other B-cell malignancies. The initial approval of ibrutinib was received on 13 November 2013 by the United States Food and Drug Administration for the treatment of adult patients with MCL who have received at least 1 prior therapy. Ibrutinib has not been approved for marketing for the treatment of aggressive B cell lymphoma although Phase I trial in this setting has already been published. In Israel ibrutinib is registered for the treatment of MCL and CLL.

DETAILED DESCRIPTION:
This is a phase II single arm clinical trial that is designed to test the efficacy of ibrutinib in combination with BR in relapsed aB-NHL either as third line post ASCT or as second or third line in non-transplant eligible patients. Patients will be referred for this study from all medical centers in Israel through the Israeli Lymphoma Working Group, but will be treated only in Chaim Sheba Medical center.

The study will include a Screening Phase, Treatment Phase, and Post- treatment Follow-up Phase.

Subject eligibility will be determined up to 30 days prior to therapy initiation. The treatment Phase will extend from cycle 1 day 1 until study drug discontinuation, either due to progression, toxicity, or due to referral to allo- SCT.

Approximately 72 eligible subjects will be stratified by background chemotherapy treatment refractory versus relapsed disease aB-NHL histology, and number of prior lines of therapy. All subject will receive BR protocol and ibrutinib 560mg per day. Ibrutinib will be administered orally once

daily starting on cycle 1, day 1, on a continuous schedule until disease progression, referral for allo-SCT, unacceptable toxicity whichever comes first. The post-treatment Follow-up Phase will begin at the end of 6 cycles of BR. Subjects who discontinue for reasons other than disease progression must continue disease evaluations.

The Post-treatment Follow-up Phase will continue until death, loss to follow up, consent withdrawal, or study end, whichever occurs first.

Assessment of tumor response and progression will be conducted in accordance with the Lugano criteria for Malignant Lymphoma. The investigator will evaluate sites of disease by radiological imaging, physical examination, or other procedures as necessary. The primary efficacy analysis of ORR will be based on investigator assessment.

At each site visit, subjects will be evaluated for toxicity. Safety evaluations will include adverse event monitoring, physical examinations, concomitant medication usage, and clinical laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over the age of 18.
2. Histologically confirmed DLBCL, Transformed low grade lymphoma to DLBCL, primary mediastinal B cell lymphoma or unclassifiable lymphoma between DLBCL and Burkitt Lymphoma, either in first or second relapse/progression in patients who are not candidates for ASCT or in second relapse/progression post ASCT (as first salvage therapy following relapse/progression post ASCT).
3. Pathology must be confirmed by a local hemato-pathologist. Patients with pathology sample over 1 year old will have to undergo a new diagnostic biopsy.
4. At least 1 prior line of therapy with rituximab containing regimen.
5. At least 1 site of measurable disease according to the Lugano criteria [1]
6. Hematology laboratory values must be within the following limits:

   1. Absolute neutrophil count (ANC)≥1000/mm3 independent of growth factor support
   2. Platelets ≥100,000/mm3 or ≥50,000/mm3 if bone marrow involvement independent of transfusion support in either situation.
7. Biochemical values within the following limits:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN unless the increase is due to Gilbert's syndrome or of non-hepatic origin
   3. Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft-Gault) ≥ 40 mL/min/1.73m2
8. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
9. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study.
10. ECOG performance status 0-2.
11. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

Prior chemotherapy radiotherapy or major surgery within 4 weeks of cycle 1 day 1.

2. Previous treatment with either bendamustine or Ibrutinib. 3. Prior allogeneic stem cell transplantation. 4. Known central nervous system lymphoma. 5. History of stroke or intracranial hemorrhage within 6 months prior to randomization.

6. Requires anticoagulation with warfarin or equivalent vitamin K antagonists. 7. Requires treatment with strong CYP3A inhibitors. 8. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.

9. Vaccinated with live, attenuated vaccines within 4 weeks of randomization. 10. Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Hbcore positive HBs negative patients will be eligible but will need to be treated with lamivudine 100 mg/day throughout the treatment phase and 6 months after it.

11. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

12. Diagnosed or treated for malignancy other than DLBCL, except:

1. Malignancy treated with curative intent and with no known active disease present for 3 years before randomization
2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
3. Adequately treated carcinoma in situ without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) of the combination of ibrutinib, bendamustine and rituximab (IBR) | 5 years
  ORR is defined as the proportion of patients having at least partial repose (PR) in interim imaging or end of chemo-immunotherapy.

SECONDARY OUTCOMES:
progression free survival (PFS) | 5 years
overall survival (OS) | 5 years
duration of response. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MEIRAV KEDMI, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Dr. Meirav Kedmi, Ramat Gan
  - Sheba medical organization, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kedmi M, Ribakovsy E, Benjamini O, Schiby G, Barshack I, Raskin S, Eshet Y, Mehr R, Horowitz N, Gurion R, Goldschmidt N, Perry C, Levi I, Aviv A, Herzog-Tzarfati K, Nagler A, Avigdor A. Ibrutinib With Bendamustine and Rituximab for Treatment of Patients With Relapsed/Refractory Aggressive B-Cell Lymphoma. Hematol Oncol. 2024 Nov;42(6):e70001. doi: 10.1002/hon.70001. PMID 39572395